CLINICAL TRIAL: NCT00002745
Title: PHASE II STUDY OF 9-AMINOCAMPTOTHECIN (9-AC/DMA, NSC# 603071) IN PREVIOUSLY TREATED HODGKIN'S DISEASE AND NON-HODGKIN'S LYMPHOMA: IWF GRADES A-H
Brief Title: Aminocamptothecin in Treating Patients With Refractory or Recurrent Hodgkin's Disease or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02791; U10CA031946 (NIH); CLB-9551; CDR0000064666 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aminocamptothecin (Experimental): aminocamptothecin
  Interventions: Drug: aminocamptothecin

INTERVENTIONS:
Drug: aminocamptothecin — 850 micrograms/square meter/day (total dose 2550 micrograms/square meter) via central venous catheter using infusion pump over 72 hours + one cycle Cycle repeated every 14 days for minimum of 6 cycles if partial or complete response

SUMMARY:
Phase II trial to study the effectiveness of aminocamptothecin in treating patients who have refractory or recurrent Hodgkin's disease or non-Hodgkin's lymphoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the response rate and duration of response to aminocamptothecin (9-AC) in patients with refractory or relapsed Hodgkin's disease or non-Hodgkin's lymphoma.

II. Assess the toxicity of 9-AC in these patients. III. Validate a preliminary pharmacodynamic model relating total 9-AC concentration, albumin, and bilirubin to toxicity.

IV. Determine whether 9-AC concentrations correlate with response.

OUTLINE: Patients are stratified by disease histology (International Working Formulation (IWF) A-C vs IWF D-F) and center.

Patients receive aminocamptothecin IV continuously on days 1-3. Treatment repeats every 2 weeks for a minimum of 3 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease, partial response (PR), or complete response (CR) may receive 2 additional courses past best response (minimum of 6 courses if PR or CR). Patients are followed every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically documented Hodgkin's disease (closed to accrual 4/15/2000) OR
* Histologically documented non-Hodgkin's lymphoma (NHL) of one of the following International Working Formulation (IWF) histologies:

  * Small lymphocytic (absolute lymphocyte count less than 5,000)
  * IWF A Follicular, predominantly small cleaved cell
  * IWF B Follicular mixed
  * IWF C Follicular large cell
  * IWF D* Diffuse small cleaved cell
  * IWF E* Diffuse mixed
  * IWF F* Diffuse large cell
  * IWF G* Large cell, immunoblastic
  * IWF H* * Accrual of patients with these diagnoses closed 4/15/2000
* Pathology review required within 60 days of registration
* Refractory to or relapsed after prior chemotherapy as follows:

  * Low-grade NHL (IWF A-C): 1 or 2 prior therapies
  * Intermediate-grade NHL (IWF D-H): 1 prior therapy (stratum closed 4/15/2000)
  * Hodgkin's disease: 1 or 2 prior therapies (stratum closed 4/15/2000)
* Treatment with the same drugs on 2 different schedules considered 1 therapy
* Measurable disease by physical exam or imaging studies
* Mass larger than 1 x 1 cm
* Documented progression required of previously irradiated lesions
* The following are not considered measurable:

  * Ascites or pleural effusion
  * Bone marrow involvement
  * Positive barium studies
  * Bony disease (lytic lesions noted)
  * No mantle cell or transformed lymphoma
  * No parenchymal or leptomeningeal CNS disease
* A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: CALGB 0-2
* Unless hypersplenism or biopsy-proven bone marrow involvement:

  * Absolute granulocyte count at least 1,500/mm3
  * Platelet count at least 100,000/mm3
* Bilirubin normal
* AST no greater than 4 times normal
* Creatinine normal
* No suspected HIV infection
* No second malignancy within past 5 years except:

  * Curatively treated carcinoma of the cervix
  * Curatively treated basal cell skin cancer
  * No uncontrolled infection or other serious medical condition
  * No psychiatric condition that precludes informed consent
  * Not pregnant or nursing
  * Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior allogeneic or autologous bone marrow transplant
* More than 3 weeks since chemotherapy (6 weeks since nitrosoureas, melphalan, or mitomycin)
* No prior camptothecin
* More than 3 weeks since radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1996-04; Primary Completion 2003-04 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Response | 2 years post treatment

SECONDARY OUTCOMES:
Toxicity | day 1 of each cycle
9-AC/DMA concentrations | Pre-treatment cycle 1 and just prior to completion of cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L. Bartlett, MD, Study Chair — Washington University Siteman Cancer Center
Locations (5):
- United States (5):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Cooper Cancer Institute, Camden, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey

REFERENCES:
- [Result] Bartlett NL, Johnson JL, Wagner-Johnston N, Ratain MJ, Peterson BA; Cancer and Leukemia Group B. Phase II study of 9-aminocamptothecin in previously treated lymphomas: results of Cancer and Leukemia Group B 9551. Cancer Chemother Pharmacol. 2009 Apr;63(5):793-8. doi: 10.1007/s00280-008-0803-x. Epub 2008 Jul 23. PMID 18648813